CLINICAL TRIAL: NCT04477954
Title: Hyperbaric Oxygen as an Adjuvant Treatment for Patients With Covid-19 Severe Hypoxemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigators and Ethic Committee endorsed early suspension of the protocol because of superiority and safety. For the interim analysys, the statistical methodology presented by Pocock was followed.
Sponsor: Asociación Argentina de Medicina Hiperbárica e Investigación (Other)
Collaborators: Hospital de Infecciosas Francisco Javier Muniz (Other Government); Hospital General de Agudos D. F. Santojanni (Unknown); Hospital Central de San Isidro Dr. Melchor Angel Posse (Unknown)
Responsible Party: Principal Investigator, Mariana Cannellotto, President, Asociación Argentina de Medicina Hiperbárica e Investigación
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAMHEI2020-1
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: Hyperbaric Oxygen; Covid-19; Hypoxemia; Sars-CoV2; Hyperbaric Chamber
MeSH Terms: conditions — COVID-19; Hypoxia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental HBOT (Experimental): Treatment (device). Patients will receive 90 minutes of hyperbaric oxygen at 1,45 ATA in a Revitalair430 hyperbaric chamber, and then they will continue with standard care and normobaric oxygen.
  Interventions: Combination Product: Hyperbaric Oxygen
- Standard care (No Intervention)

INTERVENTIONS:
Combination Product: Hyperbaric Oxygen — Hyperbaric oxygen therapy (HBOT): inhalation of pressurized oxygen through a hyperbaric chamber (Revitalair430)
  Other Names: HBOT
  Arms: Experimental HBOT

SUMMARY:
The severity of COVID-19 is related to the level of hypoxemia, respiratory failure, how long it lasts and how refractory it is at increasing concentrations of inspired oxygen. The inability to perform hematosis due to edema that occurs from acute inflammation could be attenuated by the administration of hyperbaric oxygen (HBO). Recently, it has been reported benefits in this matter in patients with SARS-CoV-2 hypoxemic pneumonia in China; where the administration of repeated HBO sessions decreased the need for mechanical ventilation (MV) in patients admitted to the Intensive Care Unit due to COVID-19. Hyperbaric oxygen is capable of increasing drastically the amount of dissolved oxygen in the blood and maintain an adequate supply oxygen to the tissues. In addition to this, it can influence immune processes, both humoral and cellular, allowing to reduce the intensity of the response inflammatory and stimulate antioxidant defenses. HBO is considered safe and it has very few adverse events, it is a procedure approved by our authorities regulatory for several years. In the current context of the pandemic by COVID-19 and worldwide reports of mortality associated with severe cases of respiratory failure, it is essential to propose therapeutical strategies to limit or decrease respiratory compromise of severe stages by COVID-19. That is why, it is proposed to carry out this research to assess whether HBO treatment can improve the evolution of patients with COVID-19 severe hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years, all sexes.
* No previous hospitalizations in the last 6 months.
* Positive diagnostic test for COVID-19 according to the guidelines of the Argetine Ministry of Health at the time of enrollment.
* Patient in Intensive Care Unit with oxygen need: Need for continuous supply of oxygen to maintain saturation by oximetry pulse (SpO2) greater than or equal to 93% or arterial gas with PaO2 value greater than 60 mmHg

Exclusion Criteria:

* 18 years of age.
* Person unable to give consent.
* Person who refuses to participate.
* Pregnancy and lactation
* Participating in other study
* Requirement for mechanical ventilation.
* Inability to maintain prolonged sitting position (at least 2 hours)
* Subject with contraindications to HBOT (pulmonary shock, bullae, emphysema or untreated pneumothorax, severe seizures, uncontrolled hypertension, chronic obstructive disease of grade III or IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Time to normalize the oxygen requirement (oxygen dependence) | 15-30 days.
  Time to normalize the oxygen requirement: Allowing a pulse oximetry value in ambient air greater than or equal 93% and/or arterial blood gas with PaO2 value greater than 60 mmHg in ambient air.

SECONDARY OUTCOMES:
Need for Invasive Mechanical Ventilation (IMV) and / or Respiratory Distress Syndrome Acute (ARDS) | 30 days
  Number of patients who required IMV after being enrolled
Development of Acute Respiratory Distress Syndrome (ARDS) | 30 days
  Number of patients who required IMV and / or had a diagnosis of ARDS after being enrolled.
30-day mortality | 30 days
  Number of patients who died in that period since enrollment
Hypotension with vasopressor requirement | 30 days
  Number of patients with hypotension who were administered vasopressors in this period
Mortality | 45 days / 60 days / 90 days and 180 days
  Number of patients who died in that period since enrollment.

OTHER OUTCOMES:
Adverse events | 4 hours finished session
  Number of adverse events reported related to the device (Revitalair 430 hyperbaric chamber): otalgias, ear obstruction, barotrauma, significant and constant changes in blood pressure, heart rate and others

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Cannellotto, MD, Study Chair — Asociación Argentina de Medicina Hiperbárica e Investigación; Mariano Duarte, PhD, Principal Investigator — Asociación Argentina de Medicina Hiperbárica e Investigación; Liliana Jorda-Vargas, Principal Investigator — Asociación Argentina de Medicina Hiperbárica e Investigación; Fabrizio Verdini, MD, Principal Investigator — Asociación Argentina de Medicina Hiperbárica e Investigación
Locations (3):
- Argentina (3):
  - Hospital Central de San Isidro Dr. Angel Melchor Posse, San Isidro, Buenos Aires
  - Hospital de Infecciosas F. J. Muñiz, Buenos Aires, Buenos Aires F.D.
  - Hospital General de Agudos D.F Santojanni, Buenos Aires, Buenos Aires F.D.

IPD SHARING:
Plan to Share IPD: No